CLINICAL TRIAL: NCT04255329
Title: Comparative Study of Two Cognitive Stimulation Approaches Using the Non-verbal Communication on People With Alzheimer's Disease and/or Related Diseases at a Moderate to Advanced Stage of Evolution
Brief Title: Non Verbal Communication and Dementia
Acronym: GEMAN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: health context of covid-19
Sponsor: University Hospital, Montpellier (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: RECHMPL18_0071
Record Dates: First submitted 2019-12-09; First posted 2020-02-05 (Actual); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Neurocognitive Disorders; Alzheimer Disease
Keywords: Non pharmacological interventions; Cognitive stimulation; Non-verbal communication; Montessori Lifestyle
MeSH Terms: conditions — Neurocognitive Disorders; Alzheimer Disease; Nonverbal Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual reading group (Other): The leader of the activity reads aloud a text to four participants seated around the table. The readen text is a normal, currently used in a everyday life support such as a journal article. Consequently it is not previously adaptated to people with cognitive impairements. After the reading phase, the leader asks the participants the questions about the content.
  Interventions: Other: Usual reading
- Montessori reading roundtable group (Other): The group counts four participants and one activity leader. Each person have the same Montessori reading roundtable book.
  Interventions: Other: Montessori reading roundtable

INTERVENTIONS:
Other: Montessori reading roundtable — Such book is written in a way to adaptate to people with cognitif and sensory impairments. Indeed, text is written in large characters and structured to not involve episodic memory. Each person read one page aloud in his turn. After the reading phase, the participants discuss the questions about their opinions and distant memories.
  Arms: Montessori reading roundtable group
Other: Usual reading — The readen text is a normal, currently used in a everyday life support such as a journal article.
  Arms: Usual reading group

SUMMARY:
Cognitive impairements in Alzheimer's and apparented disorders may lead to the decreased engagement in activities, spetially in moderate and advanced stages of evolution. The lack of stimulation for people with dementia is associated with the risk of challenging behaviors, depressives symptoms, sleeping disorders or faster cognitive deterioration. Those challenges may lead to the increased administration of pharmacological treatments, though the risks of neurleptics use in this population are currently known. In this context, non-pharacological interventions hold a significant place in dementia care.

This research focuses on cognitve stimulation activities. More precisly, our study compares two aproaches using the reading groups. The first type (" usual " reading group) is based on the principle of stimulating those cognitive functions which dicreases with the evolution of dementia. The second (Montessori reading group) approach relies on the idea to use preserved capacities in order to compensate the cognitive impariments.

The aim of our study is to compare the impact of these two non-pharmalogical interventions on non-verbal communication. The collected datas will help analyzing and understanding the internal and behavioral states of people living with dementia. Our study will also extend relfexions about cognitive stimulation groups in care institutions.

ELIGIBILITY:
Inclusion Criteria:

* 65 years and more
* Diagnosed with Alzheimer's disease and/or related disease (frontotemporal dementia, vascular dementia, multiple etiologies dementia, Lewy's Body dementia) according to DSM-IV-TR criteria (2005)
* MMSE ≤ 15
* Good reading ability assessed using Montessori Reading Test (ability to read text written in Arial 40)
* The written agreement of the patient, primary caregiver or curator or or guardian to participate in the study and to make a film about the participant.
* Patient receiving social security benefits

Exclusion Criteria:

* Previously known associated psychotic disorder
* Deafness not compensated by hearing aid
* Extrapyramidal syndrome diagnosed by a practitioner
* Tendency to daytime sleepiness (Score 6 on the Karolinska somnolence scale)
* Patient with disruptive behaviour disorders such as screaming and/or motor agitation likely to affect the smooth running of the workshop
* Subject deprived of liberty by judicial or administrative decision.
* Subject under exclusion for another research protocol.
* Presence of motor stereotypes
* Patient receiving State Medical Assistance (AME)
* Patient under Justice Safeguard
* If the patient or guardian cannot be given informed information

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02 (Estimated); Primary Completion 2021-09-27 (Actual); Study Completion 2021-09-27 (Actual)

PRIMARY OUTCOMES:
gestuality frequency | 18 months
  frequency of gestures (number of gestures observed) unrelated with the activity (item manipulations unrelated with the activity, comfort posture, self-focus gestures, look outside the interaction space) measured by ANVIL software.
gestuality duration | 18 months
  duration of gestures (duration of gestures observed in seconds) unrelated with the activity (item manipulations unrelated with the activity, comfort posture, self-focus gestures, look outside the interaction space) measured by ANVIL

SECONDARY OUTCOMES:
score in Observed Emotions Scale | 18 months
  Duration of signs of pleasure, anger, anxiety/fear, sadness and general alertness over en ten-imunt observation period in a 6 item scale : not in view ; never ; less than 16 sec. ; 16-59 sec. ; 1-5 min. ; more than 5 min. (Lawton, M.P., Van Haitsma, K. & Klapper, J.A (1999).
Score in Menorah Park Engagement Scale | 18 months
  reported participants engagement thanks to a 6 questions questionnaire : did the participant take part in the activity (yes/no) ; how long did the participant realise or comment the activity, listen/look the activity, do other things, sleep/keep eyes closed, expresse pleasure (not at all ; less than half of the time ; more than half of the time) (Camp, 2004)
Participants satisfaction | 18 months
  satisfaction self reported by participants by circle one of the tree smiley (sad ; neutral; happy)
Score in NeuroPsychiatric Inventory | 18 months
  score from 0 to 144, higher score indicated higher challenging behaviors (Sisco, F. et al., 2000).
Score in Cornell depression Scale | 18 months
  score from 0 to 38, higher score indicated higher risks of depression syndrom. (1988)

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Suzanne LEGLISE, MD, Principal Investigator — CHU of Montpellier
Locations (1):
- CHU Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No